CLINICAL TRIAL: NCT01342029
Title: Treatment With Ranolazine in Microvascular Coronary Dysfunction (MCD): Impact on Angina Myocardial Ischemia
Acronym: RWISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IN-US-259-0124 - RWISE
Record Dates: First submitted 2011-04-22; First posted 2011-04-26 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Microvascular Coronary Dysfunction (MCD)
Keywords: Microvascular Coronary Dysfunction (MCD)
MeSH Terms: interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Experimental): 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — This drug is approved by the U.S. Food and Drug Administration (FDA) for treatment of chronic angina.
  500-1,000 mg po bid for 2 weeks
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — 500-1,000 mg po bid for 2 weeks
  Arms: Placebo

SUMMARY:
This research study is designed to test the use of ranolazine in patients with angina (chest discomfort due to reduced blood supply to the heart) due to microvascular coronary dysfunction (MCD; abnormalities in the small blood vessels of the heart). This drug is approved by the U.S. Food and Drug Administration (FDA) for treatment of chronic angina. The FDA has approved this drug based on studies primarily on patients with chronic angina with major blockages of the arteries.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo- controlled, and cross-over clinical trial. 147 subjects will be enrolled at two clinical sites, with projected 9-10% dropout and anticipated 134 completed subjects. To maintain blinding of the investigators, the study randomization table will be kept in Pharmacy Service. The sponsor will ship the study drug directly to the Pharmacy Service. The pharmacy service will also be responsible for dispersing the study drug.

There are 4 study visits (2 visits in each study period) in this study. Subjects will be in this study for about 6 weeks from Week 0 - baseline visit to Week 6 - exit visit. Besides the procedure of study medication mentioned above, other study procedures include informed consent, physical exam, questionnaires, EKG for safety assessment, blood collection for laboratory testing, cardiac MRI, and follow-up events. In sum, participants will be asked to undergo 2 cardiac MRI's and fill out questionnaires 4 times. They will be asked to participate for 6 weeks with two 2-week courses (with a treatment window period of 5 days), one with ranolazine and the other with placebo (without knowing which they are taking). There is a 2-week washout period between treatments. The participants will otherwise remain on all their usual medications. The physicians will also be blinded to which medication the subject is receiving.

Participation in this study will be approximately 6 weeks, which consists of two 2-week study periods and in between a 2-week washout period:

1. During the first 2-week period: Subjects will be randomized to first receive either the ranolazine or a placebo pill (sugar pill with no active medicine). Subjects will take the extended-release ranolazine or a placebo pill for a total of 2 weeks. Subjects will take 500 mg twice daily for the first 1 week and then 1000 mg twice daily for an additional 1 week. Subjects who are unable to take the higher dose due to side effects will remain on 500 mg twice daily for the entire study period. After the 2 weeks, the participant will have a Cardiac MRI and complete study questionnaires. These tools will allow us to evaluate if the participant is doing better on the medication.
2. 2-week washout period: Subject will then be asked to go 2 weeks without any study medication (ranolazine or placebo).
3. During the second 2-week period: Subject will then be given either extended release ranolazine or placebo depending on which was received the first time for a total of 2 weeks. Subjects will take 500 mg twice daily for the first 1 week and then 1000 mg twice daily for an additional 1 week. Subjects who are unable to take the higher dose due to side effects will remain on 500 mg twice daily for entire study period. This 2-week period will again be followed by a final Cardiac MRI and questionnaire completion.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age >18 from diverse racial/ethnic groups;
2. Competent to give informed consent;
3. Patients with chronic angina or its equivalent;
4. Coronary angiogram revealing MCD with no obstructive CAD (epicardial coronary stenosis <50% luminal diameter stenosis);
5. Left ventricular ejection fraction > or = 45%;
6. Objective evidence of ischemia by noninvasive methods such as exercise stress test, stress Echo, MRI, or SPECT;
7. Patients with 10% myocardial ischemia by Cardiac magnetic resonance imaging (CMRI) myocardial perfusion reserve index ≤ 2.0 or abnormal coronary reactivity testing (CFR < 2.5, or ACH response of no dilation or constriction, determined by local site read).

Exclusion Criteria:

1. Acute coronary syndrome (defined by WHO), cardiogenic shock or requiring inotropic or intra-aortic balloon support;
2. Planned percutaneous coronary intervention or CABG or established obstructive CAD with ischemia eligible for revascularization, acute MI;
3. Prior non-cardiac illness with an estimated life expectancy <4 years;
4. Unable to give informed consent;
5. Allergy or contra-indication to CMRI testing, including renal failure, claustrophobia, and asthma, uncontrolled moderate hypertension (sitting blood pressure >160/95mmHg with measurements recorded on at least 2 occasions), conditions likely to influence outcomes: Severe lung, creatinine >1.8 or CrCl ≤ 50ml/min) or hepatic disease;
6. Surgically uncorrected significant congenital or valvular heart disease and other disease likely to be fatal or require frequent hospitalization within the next six months;
7. Adherence or retention reasons;
8. Unwilling to complete follow-up evaluation including repeat testing, documented obstructive hypertrophic cardiomyopathy;
9. Aortic stenosis (valve area <1.5cm);
10. LV dysfunction (ejection fraction ≤35%);
11. History of significant cocaine or amphetamine abuse;
12. Taking potent CYP3A4 inhibitors (ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir);
13. Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - 127 S. San Vicente Blvd, Suite A9303, Los Angeles, California
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rambarat CA, Elgendy IY, Handberg EM, Bairey Merz CN, Wei J, Minissian MB, Nelson MD, Thomson LEJ, Berman DS, Shaw LJ, Cook-Wiens G, Pepine CJ. Late sodium channel blockade improves angina and myocardial perfusion in patients with severe coronary microvascular dysfunction: Women's Ischemia Syndrome Evaluation-Coronary Vascular Dysfunction ancillary study. Int J Cardiol. 2019 Feb 1;276:8-13. doi: 10.1016/j.ijcard.2018.09.081. Epub 2018 Sep 26. PMID 30293664
- [Derived] Birkeland K, Khandwalla RM, Kedan I, Shufelt CL, Mehta PK, Minissian MB, Wei J, Handberg EM, Thomson LE, Berman DS, Petersen JW, Anderson RD, Cook-Wiens G, Pepine CJ, Bairey Merz CN. Daily Activity Measured With Wearable Technology as a Novel Measurement of Treatment Effect in Patients With Coronary Microvascular Dysfunction: Substudy of a Randomized Controlled Crossover Trial. JMIR Res Protoc. 2017 Dec 20;6(12):e255. doi: 10.2196/resprot.8057. PMID 29263019
- [Derived] Bairey Merz CN, Handberg EM, Shufelt CL, Mehta PK, Minissian MB, Wei J, Thomson LE, Berman DS, Shaw LJ, Petersen JW, Brown GH, Anderson RD, Shuster JJ, Cook-Wiens G, Rogatko A, Pepine CJ. A randomized, placebo-controlled trial of late Na current inhibition (ranolazine) in coronary microvascular dysfunction (CMD): impact on angina and myocardial perfusion reserve. Eur Heart J. 2016 May 14;37(19):1504-13. doi: 10.1093/eurheartj/ehv647. Epub 2015 Nov 27. PMID 26614823

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranolazine First, Then Placebo: 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Ranolazine: This drug is approved by the U.S. Food and Drug Administration (FDA) for treatment of chronic angina.
  500-1,000 mg po bid for 2 weeks
- Placebo First, Then Ranolazine: 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Placebo: 500-1,000 mg po bid for 2 weeks
Period: Period 1
Arm/Group | Ranolazine First, Then Placebo | Placebo First, Then Ranolazine
Started | 70 | 72
Dropout | 3 | 1
Completed | 67 | 71
Not Completed | 3 | 1
Period: Washout
Arm/Group | Ranolazine First, Then Placebo | Placebo First, Then Ranolazine
Started | 67 | 71
Completed | 67 | 67
Not Completed | 0 | 4
Period: Period 2
Arm/Group | Ranolazine First, Then Placebo | Placebo First, Then Ranolazine
Started | 67 | 67
Dropout | 2 | 0
Completed | 65 | 67
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Total 10 dropout (4 dropout during period 1, 4 dropout during washout, 2 dropout during period 2)
Groups:
- Ranolazine/Placebo: 147 subjects will be enrolled at two clinical sites, with projected 9-10% dropout and anticipated 134 completed subjects.
  For Ranolazine first group, subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  For Placebo first group, subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
Arm/Group | Ranolazine/Placebo
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 142
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Seattle Angina Questionnaire (SAQ)
Description: Questionnaires will be completed (SAQ - Seattle Angina Questionnaire) at the end of each treatment period.
  The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item questionnaire, a cardiac disease-related quality-of-life measure. The SAQ is well validated and sensitive to clinical changes. It has five subscales: physical limitation, angina stability, angina frequency, treatment satisfaction, and quality of life. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life. A change of 10 points in any of the subscales is considered to be clinically important.
Time Frame: 2 weeks (first intervention) and 6 weeks (second intervention)
Population: Not all participants answered every question in the SAQ, thus the numbers are different for each question.
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Ranolazine: 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Ranolazine: This drug is approved by the U.S. Food and Drug Administration (FDA) for treatment of chronic angina.
  500-1,000 mg po bid for 2 weeks
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 128 | 128
Units on scale
  Physical Limitation: number analyzed (Participants) | 123 | 120
  Physical Limitation | 68.09 (23.34) | 66.7 (23.34)
  Angina Stability | 58.4 (26.11) | 51.17 (27.68)
  Angina Frequency | 63.91 (26.09) | 62.73 (25.95)
  Treatment Satisfaction: number analyzed (Participants) | 127 | 128
  Treatment Satisfaction | 74.16 (21.23) | 74.17 (21.08)
  Quality of Life | 56.05 (23.09) | 54.17 (23.31)
  SAQ Overall | 62.49 (19.32) | 60.97 (20.11)

2. Secondary Outcome: Cardiac Magnetic Resonance (CMRs)
Description: Cardiac Magnetic Resonance (CMRs) (CMR 1 and CMR 2) end of the 2nd week of treatment 1 and treatment 2 respectively, 4 hours after the morning dose of study drug was performed to measure myocardial perfusion reserve index.
  Myocardial perfusion reserve index (MPRI) was assessed using the first-pass perfusion intensity curves during stress and rest cardiac magnetic resonance imaging. First-pass perfusion images were analysed using CAAS MRV CMRI analysis software Version 3.3 (Pie Medical Imaging B.V., Maastricht, the Netherlands). Global MPRI was calculated as the ratio of stress/rest relative perfusion upslope, corrected for LV cavity upslope.
  Higher MPRI represents better myocardial perfusion reserve. Since MPRI is an index, there is no unit.
Time Frame: 2 weeks (first intervention) and 6 weeks (second intervention)
Population: Out of 142 randomized, there were 10 dropouts and 4 missing treatment periods. Therefore 128 was included in analysis
Measure: Mean (Standard Deviation); unit: myocardial perfusion reserve index
Groups:
- Ranolazine: 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo basel...
- Placebo: 147 subjects with projected 9-10% dropout
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 128 | 128
myocardial perfusion reserve index | 1.98 (0.46) | 1.96 (0.42)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The SAEs are based on the publication which represent all SAEs throughout the study.
Groups:
- Ranolazine; Placebo: 147 subjects, with projected 9-10% dropout and anticipated 134 completed subjects will undergo baseline testing and then be randomized into a clinical cross-over trial of stepped dosing of ranolazine or placebo 500-1,000 mg po bid for 2 weeks with exit testing followed by cross-over to the alternate ranolazine or placebo and repeat exit testing.
  Ranolazine: This drug is approved by the U.S. Food and Drug Administration (FDA) for treatment of chronic angina.
  500-1,000 mg po bid for 2 weeks Placebo: 500-1,000 mg po bid for 2 weeks
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 14/142 | 11/142
Serious Adverse Events (participants affected / at risk) | 6/142 | 1/142
Other Adverse Events (participants affected / at risk) | 8/142 | 10/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ranolazine (N=142) | Placebo (N=142)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0) — Hospitalization
Bronchospasm (Cardiac disorders) | 1/1 (1) | 0 (0)
Chest pain, dizziness, and pre-syncope (Cardiac disorders) | 2 (2) | 0 (0)
syncope (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) — washout
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Placebo washout
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=142) | Placebo (N=142)
Nausea and dizziness (General disorders) | 3 (3) | 0 (0)
Arm shaking (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (General disorders) | 1 (1) | 0 (0)
Renal change (Endocrine disorders) | 1 (1) | 0 (0)
Throat pain, swelling and tightness (General disorders) | 1 (1) | 1 (1)
Rectocele (Endocrine disorders) | 0 (0) | 1 (1)
cough (General disorders) | 0 (0) | 1 (1)
Sinus infection (Cardiac disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 4 (4)
Excessive Sweating (Cardiac disorders) | 1 (1) | 0 (0)
Hematemesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations and Afib (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No